CLINICAL TRIAL: NCT04995133
Title: Pharmacokinetic/Pharmacodynamic Aspects of Colistin Intravenous Administration in Critically Ill Patients Suffering From Hospital Infections Caused by Multi-antibiotic-resistant Germs and Receiving Continuous Renal Replacement Therapy.
Brief Title: Colistin Intravenous Administration in Critically Ill Patients Suffering From Hospital Infections Caused by Multi-antibiotic-resistant Germs.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, NAVARRA PIERLUIGI, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3946
Record Dates: First submitted 2021-07-23; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Hospital Infection; Multi-antibiotic Resistance; Critically Ill
Keywords: Colistin
MeSH Terms: conditions — Cross Infection; Critical Illness | interventions — Colistin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colistin Arm (Experimental): Intravenous administration of 6.75 x 106 Units Colistin for 30 minutes
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Colistin — intravenous administration

SUMMARY:
Colistin is an antibiotic active against several classes of multi-resistant gram-negative bacteria; the drug should be used in high doses in patients on continuous renal replacement therapy, since the drug is eliminated through the dialysis filter.

This is an Open-label, Phase 4, interventional, prospective, single-center pilot study aimed to analyze the concentrations of colistin in plasma and ultrafiltrate by liquid chromatography/mass spectrometry, in 20 critically ill patients admitted to intensive care and suffering from severe infections by multi-resistant bacteria, who receive continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Infection where the involvement of MDR germs is documented or highly probable
* Continuous renal replacement therapy
* Acute renal failure, stage III of the 2012 KDIGO classification
* Half-life of the continuous renal replacement therapy filter less than 48 hours.

Exclusion Criteria:

* State of pregnancy or breastfeeding, or patients expecting to conceive children within the projected duration of the study, starting with the screening through 30 days after the last dose of IMP treatment
* Patients with a positive urine pregnancy test within 72 hours prior to study drug treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Women of childbearing potential
* Refusal of informed consent
* Known hypersensitivity to polymyxins and to excipients
* Clinical condition with high probability of death, according to Symplified Acute Physiology Score (SAPS II)
* Partial maintenance of renal function, defined by stages I and II of the 2012 KDIGO classification.
* Renal replacement therapy filter other than AN69 ST 150
* Prior systemic treatments with any investigational agents within 4 weeks prior to the inclusion in the trial
* Any other clinical condition that, in the opinion of the investigator, makes the patient unfit for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0-12 hours
  Colistin A and B misuration in the plasma and in the pre-post filter.
Peak plasma concentration | 0-12 hours
  Colistin A and B misuration in the plasma
Half-life | 0-12 hours
  Colistin A and B misuration in the plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico A.Gemelli IRCSS, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Pascale G, Lisi L, Cutuli SL, Marinozzi C, Palladini A, Ferrando ES, Tanzarella ES, Lombardi G, Grieco DL, Caroli A, Xhemalaj R, Cascarano L, Ciotti GMP, Sandroni C, Sanguinetti M, Navarra P, Antonelli M. High-dose colistin pharmacokinetics in critically ill patients receiving continuous renal replacement therapy. Ann Intensive Care. 2024 Sep 28;14(1):152. doi: 10.1186/s13613-024-01384-1. PMID 39340688